CLINICAL TRIAL: NCT06555731
Title: Long-read Human Genome Sequencing in 72 Hours: "Ultra Rapid GEnome Sequencing"
Brief Title: Ultra Rapid GEnome Sequencing
Acronym: URGES
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/03
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Whole Genome Sequencing
Keywords: Next Generation Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteers
  Interventions: Genetic: Ultra rapid genome sequencing

INTERVENTIONS:
Genetic: Ultra rapid genome sequencing — DNA extraction from blood sample and whole genome sequencing

SUMMARY:
Next-generation sequencing (NGS) has revolutionized the field of genomics, allowing the detection of genetic abnormalities for diagnostic or therapeutic purposes. Turnaround times for exome or genome sequencing results have decreased to an average of 3 to 6 months.

An increasing number of diagnostic and therapeutic fields are benefiting from the advancements in ultra-rapid sequencing. In some situations, a shorter turnaround time may be useful for making therapeutic and/or interventional management decisions.

This study aims to explore the feasibility of very rapid whole-genome sequencing, ultra-rapid genome sequencing (URGES) in 72 hours, that could benefit patients with cancer or rare diseases.

DETAILED DESCRIPTION:
* Blood sample (5 ml)
* Extraction of genomic DNA from lymphocytes
* Ultra-rapid genome sequencing (48 hours for a whole genome), using the PromethION P2 Solo sequencer (Oxford Nanopore Technologies)
* Bioinformatics analysis of raw high-throughput sequencing data with SeqOne platform
* Medical interpretation of molecular data: NGS data must be interpreted by a multidisciplinary decision-support team to determine mutation actionability and identify potential "drivers"

ELIGIBILITY:
Inclusion Criteria:

* No known progressive or chronic diseases
* Consent for participation
* Affiliation to a social security system

Exclusion Criteria:

* Unable to understand
* Pregnant or breastfeeding women
* Subject under protection of the adults (guardianship, curators or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with no known progressive or chronic diseases
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Time (in hours) for long read human genome sequencing and data interpretation | 72 hours
  Time (in hours) to complete a long-read human genome sequencing, from the extracted DNA to the molecular and clinical results

SECONDARY OUTCOMES:
Sequencing coverage | 72 hours
  >30 X respective to refseq BED
Sequencing depth | 72 hours
  >30 X respective to refseq BED
Number of variants called appropriately or not | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Rafaël, Levallois-Perret, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No